CLINICAL TRIAL: NCT05425667
Title: Sensory System Weighting and Sensory Integration Therapy Training in Patients With Lumbar Spinal Stenosis
Brief Title: Sensory Integration Therapy Training in Patients With Lumbar Spinal Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201912150RINA
Record Dates: First submitted 2022-06-13; First posted 2022-06-21 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-03

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Lumbar spinal stenosis; Functional assessment; Center of pressure; Balance ability
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): sensory integration training exercise for improving balance and walking ability of patients with lumbar stenosis and neurological claudication.
  Interventions: Other: virtual reality walking training

INTERVENTIONS:
Other: virtual reality walking training — The sensory integration training of this project will combine virtual reality technology and balance interference treadmill, and manipulate vision, vestibular sense and proprioceptive systems as the main training goals. It is expected to train twice a week for 1 hour, for a total of 6 weeks of training , in order to improve the balance and walking ability of patients with lumbar stenosis and neurological claudication, and to promote the ability of subjects to transfer the effect to daily life after training.

SUMMARY:
Lumbar spinal stenosis is a common degenerative disease in the elderly. Patients are often accompanied by paresthesias and decreased musculoskeletal system functions, resulting in disability and increasing the burden of medical care. The balance and walking ability of such patients are affected by the compressed nerves, so it is necessary to reorganize the nerve sensory systems to compensate for the disability caused by lumbar stenosis. It is necessary to strengthen the training of sensory integration ability, but it has not been Studies have investigated which treatments or surgery can improve sensory integration in patients with lumbar stenosis. Therefore, this study will develop a clinical tool to objectively evaluate sensory integration, quantify the sensory integration ability of patients with lumbar stenosis and neurological claudication; The influence and mechanism of the balance ability.

DETAILED DESCRIPTION:
Objective 1. To develop a sensory integration assessment tool for patients with lumbar stenosis, in order to explore the distribution ratio of sensory system weights between them and healthy elders of the same age without lumbar stenosis under different balance disturbance stimuli.

Objective 2. To explore the distribution ratio of sensory system weights and long-term tracking of changes in sensory system weights in patients with lumbar stenosis and neurological claudication who received sensory integration training after spinal decompression surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 50 and 79 years old
2. Patients with lumbar stenosis and neurological claudication diagnosed according to MRI
3. Timed sit-stand-walk test greater than 9 seconds
4. Can stand independently for more than 30 seconds

Exclusion Criteria:

1. previous lumbar surgery
2. neurological disorder such as stroke or spinal cord injury
3. metabolic disease such as diabetes mellitus
4. vestibular disease such as Meniere's disease.

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Postural balance: Mean velocity | 1 year
  The postural balance measurements are performed by using a force platform. The data from the force platform is used to calculate the mean velocity (unit: cm/s).
Postural balance: Mean distance | 1 year
  The postural balance measurements are performed by using a force platform. The data from the force platform is used to calculate the mean distance (unit: cm).
Postural balance:Ｍean frequency | 1 year
  The postural balance measurements are performed by using a force platform. The data from the force platform is used to calculate the mean frequency (unit: Hz).
Postural balance: Ellipse area | 1 year
  The postural balance measurements are performed by using a force platform. The data from the force platform is used to calculate 95% confidence ellipse area (unit: cm^2).
Functional assessment: Walking speed | 1 year
  Functional assessment is a process that allows for the identification of disability. The data from the functional assessment is used to calculate walking speed (unit: m/s).
Functional assessment: Walking distance | 1 year
  Functional assessment is a process that allows for the identification of disability. The data from the functional assessment is used to calculate walking distance (unit: m)
Functional assessment: Duration | 1 year
  Functional assessment is a process that allows for the identification of disability. The data from the functional assessment is used to calculate the duration it took to complete the test (unit: s).
Muscle activities | 1 year
  Electromyography is a technique for evaluating and recording muscle activity. The data from electromyography is used to calculate a normalized value (unit: ratio).
Kinematic variables: Joint angles | 1 year
  A motion capture system is used to measure the joint kinematics. The data is used to calculate joint angles (unit: degree).
Kinematic variables: Center of mass | 1 year
  A motion capture system is used to measure the joint kinematics. The data is used to calculate the displacement of the center of mass (unit: cm).

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Hsu, Ph.D, Principal Investigator — National Taiwan Unversity
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No